CLINICAL TRIAL: NCT01689948
Title: Alzheimer Disease : Rehabilitation's Intervention at Home. A Preliminary Pilot Study.
Brief Title: Alzheimer Disease : Rehabilitation's Intervention at Home
Acronym: pré MATAPA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties of recruitment
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC12_0080
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Alzheimer's Disease
Keywords: Home care, rehabilitation therapy, Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home rehabilitation therapy (Experimental): 12 weekly sessions of Home rehabilitation therapy
  Interventions: Behavioral: Home rehabilitation therapy

INTERVENTIONS:
Behavioral: Home rehabilitation therapy — 12 sessions of home rehabilitation therapy

SUMMARY:
Alzheimer's disease (AD) is the most common cause of dementia among elderly patients. By its prevalence and its medical and social consequences, AD represents a dual challenge to public health and society. The elderly want to stay in their homes even when their lives are altered by a chronic progressive disease. Their caregivers claim in turn a support at home. But this desire is questioned because of the characteristics of the disease, e.g. the altered relational function by the cognitive impairment and the behavioural disorders associated.

Outpatients non-drug therapies represent a potential support that adapts to patient with an AD or mixed dementia, especially in their milder forms.

The aim of the study is to evaluate the feasibility of a weekly rehabilitation's intervention at home and its acceptability by both the patient and the caregiver.

The study of its efficiency in terms of autonomy will be the next step.

DETAILED DESCRIPTION:
The protocol is based on weekly rehabilitation's intervention at home. All home visits and assessments of the patient and his caregiver will be made by the rehabilitation's therapist himself.

Twelve weekly interventions at home are planed. The first five are needed to define a realistic and achievable goal of treatment which is accepted by the dyad and the therapist. The following seven interventions will achieve this goal by rehabilitation's intervention (e.g. occupational therapy, psychomotor approach).

Four filmed sessions for dyad's assessment are planned (at inclusion, at weeks 5 and 12 after inclusion and 3 months after the last intervention).

ELIGIBILITY:
Patient's inclusion criteria:

* Aged 65 and over
* AD or mixed dementia (DSM IV TR criteria), documented by a neuropsychological assessment and a brain imaging
* Living at home
* Having a caregiver (more than 2 visits per week)
* Agreement for the study

Caregiver's inclusion criteria :

* More than 2 patient's visits per week
* Agreement for the study

Patient's exclusion criteria:

* Life expectancy less than 1 year
* Guardianship
* Already having a rehabilitation program's therapy
* Participation in a pharmacological study

Caregiver's exclusion criteria:

- Medical condition requiring regular care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the mean scores of Instrumental Activities of Daily Living (IADL) | 27 weeks
  The main objective is to compare the mean scores of Instrumental Activities of Daily Living (IADL) observed at inclusion (day 0) with those observed 27 weeks later (meaning 3 months after the last of the twelfth weekly session of at home rehabilitation therapy).

SECONDARY OUTCOMES:
Evaluation of the mean scores of Instrumental Activities of Daily Living (IADL) | 5 weeks
  This objective is to compare the mean scores of Instrumental Activities of Daily Living (IADL) observed at inclusion (day 0) with those observed 5 weeks later (meaning after the fifth weekly session of at home rehabilitation therapy).
Evaluation of the mean scores of Instrumental Activities of Daily Living (IADL) | 13 weeks
  This objective is to compare the mean scores of Instrumental Activities of Daily Living (IADL) observed at inclusion (day 0) with those observed 13 weeks later (meaning after the twelfth weekly session of at home rehabilitation therapy).
Evaluation of the mean scores of Neuro Psychiatric Inventory (NPI) | 27 weeks
  This objective is to compare the mean scores of Neuro Psychiatric Inventory(NPI) observed at inclusion (day 0) with those observed 27 weeks later (meaning 3 months after the last of the twelfth weekly session of at home rehabilitation therapy).
Evaluation of the mean scores of Neuro Psychiatric Inventory (NPI) | 5 weeks
  This objective is to compare the mean scores of Neuro Psychiatric Inventory(NPI) observed at inclusion (day 0) with those observed 5 weeks later (meaning after the last of the fifth weekly session of at home rehabilitation therapy).
Evaluation of the mean scores of Neuro Psychiatric Inventory (NPI) | 13 weeks
  This objective is to compare the mean scores of Neuro Psychiatric Inventory(NPI) observed at inclusion (day 0) with those observed 12 weeks later (meaning after the last of the twelfth weekly session of at home rehabilitation therapy).
Evaluation of the mean scores of Zarit's scale (caregiver burden) | 13 weeks
  This objective is to compare the mean scores of Zarit's scale observed at inclusion (day 0) with those observed 13 weeks later (meaning after the twelfth weekly session of at home rehabilitation therapy).
Evaluation of the mean scores of Zarit's scale (caregiver burden) | 27 weeks
  This objective is to compare the mean scores of Zarit's scale observed at inclusion (day 0) with those observed 27 weeks later (meaning 3 months after the last of the twelfth weekly session of at home rehabilitation therapy).
Evaluation of the mean scores of Zarit's scale (caregiver burden) | 5 weeks
  This objective is to compare the mean scores of Zarit's scale observed at inclusion (day 0) with those observed 5 weeks later (meaning after the last of the fifth weekly session of at home rehabilitation therapy).
Alcohol consumption for the patient and the caregiver | 27 weeks
  This objective is to compare the alcohol consumption for the patient and the caregiver observed at inclusion (day 0) with those observed 27 weeks later (meaning 3 months after the last of the twelfth weekly session of at home rehabilitation therapy).
Evaluation of the mean scores of Mini Mental State Examination (MMSE)(meaning evaluation of patient's cognitive impairment) | 27 weeks
  This objective is to compare the mean scores of Mini Mental State Examination (MMSE) observed at inclusion (day 0) with those observed 27 weeks later (meaning 3 months after the last of the twelfth weekly session of at home rehabilitation therapy).
Evaluation of the mean scores of Goal Attainment scales (GAS) (meaning evaluation of the satisfaction of the patient and of her/his caregiver) | 27 weeks
  This objective is to compare the mean scores of Goal Attainment Scales (GAS) observed at inclusion (day 0) with those observed 27 weeks later (meaning 3 months after the last of the twelfth weekly session of at home rehabilitation therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Berrut, Pr, Principal Investigator — Bellier Hospital, CHU of Nantes
Locations (1):
- Bellier Hospital, CHU of Nantes, Nantes, France